CLINICAL TRIAL: NCT00010608
Title: Clinical Trial of Meditation for Cardiovascular Disease in Older Black Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: Howard University (Other); Morehouse College of Medicine (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P50AT000082-01P2 (NIH); P50AT000082-01 (NIH); P50AT000082-02 (NIH)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Cardiovascular Diseases
Keywords: CVD
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcendental Meditation program (Experimental): A mental technique for stress reduction which is natural, easy and effortless and is practiced sitting in a chair with eyes closed for 20 minutes twice a day.
  Interventions: Behavioral: Transcendental Meditation
- Health Education (Active Comparator): A lifestyle modification program for improving diet, exercise, salt intake and substance use.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Transcendental Meditation — a mantra meditation technique which originated from the Vedic tradition of India. It is practiced from 20 minutes twice a day sitting comfortably in a chair with eyes closed.
  Arms: Transcendental Meditation program
Behavioral: Health Education — didactic education classes for lifestyle modification through diet, exercise, substance use control, and salt intake
  Arms: Health Education

SUMMARY:
The purpose of this study is to evaluate the effectiveness of meditation in preventing of atherosclerotic cardiovascular disease (CVD) in postmenopausal, older African American women.

DETAILED DESCRIPTION:
Older African American women suffer from disproportionately high rates of cardiovascular (CVD) morbidity and mortality compared to white Americans. Numerous controlled studies suggest that this disparity is associated with chronic psychosocial and environmental stress. Research indicates that Transcendental Meditation (TM) may result in significant improvements in CVD risk factors in this high risk population.

Participants in this study will be randomly assigned to either active stress reduction with TM or health education control, both in addition to usual medical care, for 12 months. The primary outcome will be carotid artery atherosclerosis (IMT) measured non-invasively by quantitative B-mode ultrasonography. Secondary measures will include traditional CVD risk factors (blood pressure, serum glucose and insulin levels, obesity, and sedentary lifestyle), stress-related neurohormones (catecholamine metabolite and cortisol), psychosocial stress, and quality of life. The results of this trial will yield valuable new knowledge for the prevention of CVD through a CAM intervention in high risk older African American women.

ELIGIBILITY:
Inclusion Criteria:

* African American, self-identified
* Coronary artery disease (CAD/CHD) defined by laboratory examination or documented clinical history of: a)myocardial infarction; b) coronary revascularization procedure--CABG, PTCA; c) coronary angiography--at least one coronary artery with >50% stenosis
* Informed consent
* Written Permission of participant's referring physician

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 1999-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Carotid artery atherosclerosis (IMT) measured non-invasively by quantitative B-mode ultrasonography | one year

CONTACTS AND LOCATIONS:
Overall Officials: Robert H. Schneider, MD, Principal Investigator — Center for Health and Aging Studies
Locations (3):
- United States (3):
  - Howard University Medical Center, Washington D.C., District of Columbia
  - Morehouse School of Medicine, Atlanta, Georgia
  - Maharishi University of Management, Fairfield, Iowa